CLINICAL TRIAL: NCT02338596
Title: Comparison of the Outcomes of Ultra-Short Anatomic and Conventional Cementless Stems in Patients Younger Than Fifty-Five Years Old
Brief Title: Ultra-Short Anatomic and Conventional Cementless Stems Cementless Stems in Patients Younger Than Fifty-Five Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shortstem005
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Hip Replacement, Total; Osteonecrosis of Femoral Head; Coxarthrosis
MeSH Terms: conditions — Femur Head Necrosis; Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional stem (Experimental): total hip replacement operated with conventional stem (Profile; DePuy, Leeds, United Kingdom)
  Interventions: Procedure: Total hip replacement
- Ultra-Short stem (Active Comparator): total hip replacement operated with ultra-short stem (Proxima; DePuy, Leeds, United Kingdom)
  Interventions: Procedure: Total hip replacement

INTERVENTIONS:
Procedure: Total hip replacement — 1. Simultaneous bilateral sequential total hip arthroplasties under the same anesthetic.
  2. Randomization to treatment with an ultra-short or a convnetional cementless stem was accomplished with use of study numbers in sealed envelope, which were opened in the operating room before the skin incision was made.
  3. The pore size was 250㎛. A 28-mm-diameter Biolox forte ceramic femoral head (CeramTec AG, Polchingen, Germany) ) was used in all hips. A cementless cup and a 28mm internal-diameter Biolox forte ceramic liner was used in all hips in both groups.

SUMMARY:
As clinical and radiographic performance of an ultra-short anatomic cementless stem have been investigated only two randomized controlled studies, well-designed trials should aim for a thorough comparison of the outcomes of ultra-short and conventional cementless stems. The purpose of this study was to compare the outcomes of ultra-short and conventional stems in the same young patients who underwent simultaneous bilateral sequential total hip arthroplasties.

DETAILED DESCRIPTION:
Conventional cementless femoral stems are known to provide a high rate of satisfactory clinical outcomes at long-term follow-ups. However, they may have potential clinical consequences related to stress shielding, thigh pain, periprosthetic fractures, proximal/distal dimensional mismatch, an easier access pathway for wear debries and removal during revision. In an effort to reduce the risk of stress shielding, thigh pain, periprosthetic fracture, proximal/distal stem mismatch, and to facilitate removal of well fixed stem, a new ultra-short anatomic metaphyseal-fitting cementless femoral stem was developed. It was designed to provide closely mimicking the original functioning hip. The absence of the diaphyseal anchorage attempt proximal load transfer to reduce stress shielding, thigh pain and proximal distal/mismatch. Furthermore, it attempts to preservation of the femoral canal and femoral elasticity and ease of revision. The question thus arises whether it is possible to obtain strong and long-lasting fixation of the femoral component without diaphyseal anchoring.

As clinical and radiographic performances of this ultra-short stem have been investigated only in a few studies and at short-term follow-ups, it remains to be elucidated whether an ultra-short stem shows a low incidence of implant loosening, stem misalignment, intraoperative fractures and revision rate. The purpose of this randomized controlled study to compare: (1) the clinical results, including Harris hip score, thigh pain, Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index score, and patients' satisfaction; (2) radiographic results, including stress shielding, implant loosening, stem misalignment; and (3) intraoperative fractures and revision rates of cementless total hip arthroplasty using an ultra-short anatomic metaphyseal-fitting cementless femoral stem versus a conventional metaphyseal and diaphyseal fitting anatomi proximal porous-coated cementless stem in the same patients who underwent bilateral simultaneous sequential total hip arthroplasty under one anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* End stage hip arthritis

Exclusion Criteria:

* Age above 50 years old
* Inflammatory arthritis
* Coexisting foot or ankle disorder limiting walking

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2001-06; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Thigh pain | 10 year after the operation
  thigh pain,in visual analog scale 0 to 10.

SECONDARY OUTCOMES:
Harris hip score | 10 year after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, M.D., Principal Investigator — Professor